CLINICAL TRIAL: NCT00536302
Title: A Single Center, Prospective, Randomized, Placebo-Controlled, Double-Blind Pilot Clinical Trial to Evaluate the Sensitivity of Magnetic Resonance Imaging to Detect Change in Cartilage Structure and Composition in 30 Participants Diagnosed With Osteoarthritis of the Knee and Treated With Collagen Hydrolysate
Brief Title: A Placebo-Controlled Study of Collagen Hydrolysate in Subjects With Knee Osteoarthritis (OA)
Acronym: NMR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GELITA (Industry)
Responsible Party: Timothy E. McAlindon, MD, MPH - Principal Investigator, Tufts Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gelita TM 1
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Knee Osteoarthritis (OA)
Keywords: OA; Knee arthritis; Osteoarthritis; Nutritional supplement; CAM; MRI
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Collagen Hydrolysate
  Interventions: Dietary Supplement: Collagen Hydrolysate
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Collagen Hydrolysate — Collagen Hydrolysate solution 10 grams per day by mouth for 48 weeks
  Arms: 1
Dietary Supplement: Placebo — Matching placebo solution per day by mouth for 48 weeks.
  Arms: 2

SUMMARY:
This study is designed to evaluate, by MRI, knee cartilage and structure in all subjects. Half the subjects in this study will take collagen hydrolysate each day for 48 weeks and the other half of the subjects will take a placebo dose, that looks like and tastes like the collagen hydrolysate, each day for 48 weeks. MRIs will be taken at Study Weeks -1, 24, and 48.

DETAILED DESCRIPTION:
This is a single-site, double-blind, pilot study to evaluate the sensitivity of MRI to detect cartilage structure and composition in subjects taking daily oral collagen hydrolysate (a nutritional supplement) or placebo for 48 weeks. 30 subjects will be randomized to collagen hydrolysate or placebo (1:1 ratio). The goal is to evaluate, by MRI, knee cartilage and structure in all subjects. The primary functional outcome measure will be the WOMAC questionnaire and the primary pathological outcome measure will be knee cartilage structure and composition as measurements done by MRI imaging. Subjects will have contrast dGEMRIC MRIs done at Study Weeks -1, 24 and 48.

ELIGIBILITY:
Inclusion Criteria:

* age > 49 years
* chronic knee discomfort based on the affirmative response to the question "During the past 6 months, have you had any pain in the knee more than half the days of the month ?"
* WOMAC pain subscale score ≥ 1
* tibiofemoral or patellofemoral osteoarthritis on anteroposterior weight-bearing semi-flexed or lateral knee radiographs with at least one osteophyte and no significant joint-space-narrowing
* clinical examination confirming knee pain or discomfort referable to the knee joint
* prepared to refrain from use of glucosamine, chondroitin, sAME and doxycycline
* stable medication and/or supplement use

Exclusion Criteria:

* use of glucosamine, chondroitin, diacerein or doxycycline within 14 weeks prior to randomization
* serious medical conditions or impairments that, in the view of the investigator, would obstruct their participation in the trial
* individuals who are expected not to comply with the study protocol
* plan to permanently relocate from the region during the trial period
* planned knee arthroplasty in the study knee
* active pathology of confounding origin which may cause pain, extending to the knee
* pregnancy
* any contra-indication to having an MRI scan

Ages: 49 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To measure the effect of collagen hydrolysate on knee cartilage as measured by MRI. | 48 Weeks

SECONDARY OUTCOMES:
To measure knee cartilage volume over 48 weeks at three time points. | 48 Weeks
To measure and evaluate WOMAC pain subscale scores over 48 weeks. | 48 Weeks
To evaluate change in physical function tests over 48 weeks. | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E McAlindon, MD, MPH, Principal Investigator — Tufts Medical Center; Center for Arthritis and Rheumatic Diseases
Locations (1):
- Tufts Medical Center; Center for Arthritis and Rheumatic Diseases, Boston, Massachusetts, United States

REFERENCES:
- [Derived] McAlindon T, Bartnik E, S Ried J, Teichert L, Herrmann M, Flechsenhar K. Determination of serum biomarkers in osteoarthritis patients: a previous interventional imaging study revisited. J Biomed Res. 2016 Oct 17;31(1):25-30. doi: 10.7555/JBR.31.20150167. PMID 28808182